CLINICAL TRIAL: NCT06604195
Title: Effectiveness of Modified Sciatic Nerve Mobility Exercises on Hamstring Length in Collegiate Students With Hamstring Tightness - A Randomized Controlled Study.
Brief Title: Modified Sciatic Nerve Mobility Exercises on Hamstring Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-34-MAR-2023
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Hamstring Tightness
Keywords: Hamstring tightness; Neurodynamic; neural mobilization; Muscle stretching

STUDY DESIGN:
Intervention Model Description: The participants in this study are allocated in two groups, group 1 and group 2.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is blinded to the treatment allocation to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: MSNM (Experimental): The participants in this group are treated with modified sciatic nerve mobilization.
  Interventions: Procedure: Modified sciatic nerve mobility exercises
- Group 2: DHMS (Active Comparator): The participants in this group are treated with dynamic hamstring muscle stretching.
  Interventions: Procedure: Dynamic hamstring muscle stretching

INTERVENTIONS:
Procedure: Modified sciatic nerve mobility exercises — Each participant was made to lie down in a supine position on the treatment couch. The participant's leg was moved to about 30-45 degrees hip flexion with knee extension. The ankle was then moved to maximum dorsiflexion with inversion and hip internal rotation within the participant's tolerance, and this position was maintained for 30 seconds. While the therapist performed dorsiflexion with inversion and hip internal rotation in the supported straight leg raise position, the participant was instructed to actively flex the cervical spine slowly until they perceived a tolerable stretch sensation in the hamstring muscle and lower leg. The synchronous alternating movements were performed rhythmically for 10-15 repetitions. This maneuver was repeated 3 times in a single session, 3 days per week, and continued for 3 consecutive weeks.
  Arms: Group 1: MSNM
Procedure: Dynamic hamstring muscle stretching — The participant was instructed to stand straight with the unaffected foot supported on the floor and the toes pointing forward. The heel of the testing leg was placed on an 18" high step with the toes directed upwards with knee extension. Once cued, the participant was asked to flex forward at the hip while maintaining the spine in a neutral position and reaching the arms forward. The knee joint remained fully extended as the participant continued to flex the hip until a gentle stretch was felt in the posterior thigh. Once the position was achieved, the participants were asked to hold it for 20-30 seconds. The same procedure was repeated 3 times daily, 3 days a week for three consecutive weeks.
  Arms: Group 2: DHMS

SUMMARY:
This study included collegiate students with tight hamstring muscles aged between 18-23 recruited from the Gulf Medical University, Ajman, UAE to compare the effectiveness of modified sciatic nerve mobility exercises and dynamic hamstring muscle stretching (DHMS) on hamstring length in collegiate students with hamstring muscle tightness.

DETAILED DESCRIPTION:
Hamstring Muscle Tightness is a common musculoskeletal condition that affects a significant proportion of the general population, particularly among collegiate students. Among the student population, sitting for longer periods during college hours is the primary cause of HMT. Evidence suggests that stretching with a combination of manual or instrument-assisted soft tissue mobilization are effective in improving hamstring muscle flexibility among individuals with HMT. A meta-analysis demonstrated a significant improvement in knee extension ROM and straight leg raise test measures following neural mobilization treatment which support the effectiveness of neural mobilization treatment in enhancing hamstring flexibility compared to muscle inhibition and stretching techniques . Especially, neural glides and neural stretching designed to restore the overall balance in the nervous system and can increase hamstring muscle flexibility, making them valuable interventions for individuals with HMT. A study on hamstring muscle flexibility in relation leg rotation suggest that hamstring stretching is enhancing the leg rotation and hamstring lengthening. Thus, dynamic stretching targeting the nerves and muscles is warranted for the treatment of tight hamstring in the general population, especially among collegiate students. This evidence provides input for the modification of dynamic sciatic nerve stretching to improve the effects of therapeutic interventions that focus on neuromuscular flexibility, joint ROM, and pain relief. Further evidence also suggests that nerve-directed stretching is superior to muscle-directed stretching in improving hamstring tightness in healthy adults. However, the role of nerve-directed dynamic stretching with hip rotation has not been addressed by previous interventional studies. Therefore, This study compared the effects of modified sciatic-nerve mobility exercises over dynamic hamstring muscle stretching on improving the hamstring length in collegiate students with HMT to determine the most effective approach for managing this condition.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate students with hamstring muscle tightness.
* Unilateral and/or bilateral hamstring muscle tightness.
* Students from the Gulf Medical University.

Exclusion Criteria:

* History of intervertebral disc lesions and radiculopathies,
* Soft tissue injuries in the lower extremity.
* Spine surgery, lower extremity neurological complications.
* Students engaged in competitive sports.
* Students engaged in other interventional studies.
* Lower back pain from specific causes.
* Pelvic inflammatory conditions.
* Unwillingness to provide informed consent.
* Nutritional deficiencies.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Passive Knee Extension (PKE) ROM test | Baseline, post-treatment day 1, end of week 1, and week 2
  To measure the hamstring length using Passive Knee Extension (PKE) ROM test, the participant was in supine position on the plinth, the hip and knee of the lower limb to be tested kept at 90° flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Ramprasad Muthukrishnan, PhD, Study Chair — Gulf Medical University
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The data may be provided based upon request related to research purpose